CLINICAL TRIAL: NCT06989125
Title: Internet-based Versus Synchronous Cognitive Behavioural Therapy for Patients With Gambling Disorder: A Non-inferiority Randomized Controlled Trial
Brief Title: Internet-based Versus Synchronous Cognitive Behavioural Therapy for Patients With Gambling Disorder
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Aarhus University Hospital (Other)
Collaborators: University of Aarhus (Other)
Responsible Party: Principal Investigator, Lisbeth Frostholm, Professor, Aarhus University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1-10-72-145-24; DLK-2308_002 (Other Grant/Funding Number: Dansk LudomaniKomité); 2023-4552 (Other Grant/Funding Number: The Danish Ministry of the Interior and Health)
Record Dates: First submitted 2025-02-21; First posted 2025-05-25 (Actual); Last update posted 2025-05-25 (Actual); Status verified 2025-05

CONDITIONS: Gambling Disorder
Keywords: Gambling Disorder treatment; Internet-based treatment; Cognitive behavioral therapy; Non-inferiority trial; Randomized controlled trial
MeSH Terms: conditions — Gambling

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Internet-based cognitive behavioral therapy ("SpilleFri") (Experimental): Participants in this arm receive internet-based cognitive behavioral therapy via the therapist-guided online treatment platform "SpilleFri"
  Interventions: Behavioral: Internet-based cognitive behavioral therapy
- Synchronous cognitive behavioral therapy (sCBT) (Active Comparator): Participants in this arm receive traditional synchronous cognitive behavioral therapy, face-to-face or via video-connection
  Interventions: Behavioral: Synchronous cognitive behavioral therapy

INTERVENTIONS:
Behavioral: Internet-based cognitive behavioral therapy — The internet-based CBT treatment arm is delivered via the online treatment platform "SpilleFri" and consists of nine internet-delivered modules delivered over 10-12 weeks. Modules contain written assignments and multiple-choice lists, combined with psychoeducation delivered in text, illustrations, and videos. The treatment is assisted by a therapist. The therapist contact is primarily written and takes place in an embedded secured message system on the platform. Participants can use the written message function whenever they want, and the therapist will respond on a specific day each week. Further, participants are offered up to three sessions of face-to-face or video-based therapist support during the treatment, depending on their preference.
  Treatment is regarded as completed if the participant has worked actively (logged in to the module and filled in at least one interactive exercise) in the first 6 modules of the treatment program.
  Other Names: SpilleFri
  Arms: Internet-based cognitive behavioral therapy ("SpilleFri")
Behavioral: Synchronous cognitive behavioral therapy — In the sCBT condition, participants receive 9 individual sessions spread over 14-20 weeks, in a 1 to 1 format with a therapist, delivered either face-to-face or via video connection, depending on the participant's preference (there may be a mix). Treatment sessions take place weekly at the start of the course. After week 4, the aim is to have sessions at least every other week to maintain continuity in treatment. Further, participants are offered up to three additional sessions that can be included on request of participant or when therapists deem it necessary. Treatment is regarded as completed if the participant has attended 6 sessions of the treatment program.
  Other Names: Face-to-face CBT
  Arms: Synchronous cognitive behavioral therapy (sCBT)

SUMMARY:
The aim of this two-armed, randomized controlled trial is to determine if internet-based cognitive behavioural therapy (CBT) is as effective as synchronous CBT (sCBT) for treating Gambling Disorder (GD) in adults. The main question it aims to answer is: Is the effect of the internet-based CBT ("SpilleFri") non-inferior to that of synchronous CBT in reducing gambling severity?

The trial will enroll 150 patients with Gambling Disorder who will be randomized (1:1) to either the experimental condition (12 weeks' treatment with the internet-based treatment "SpilleFri") or the active control condition (18 weeks individual sCBT). The primary outcome measure will be based on self-reported GD severity (NODS).

The trial will be considered effective if SpilleFri is not clinically inferior (within a predefined non-inferiority margin) to sCBT in reducing GD severity at the primary endpoint three months after end-of-treatment.

In addition to evaluating the effectiveness of the treatments, the study will conduct an exploratory analysis of the impact of each condition on secondary outcomes (changes in gambling behavior, relationship quality, and symptoms of anxiety, depression, and emotional distress). Similarly, an exploratory analysis of process variables (gambling-related self-efficacy, maladaptive gambling cognitions, emotion regulation difficulties, and gambling urge) will be conducted across conditions and clinical subgroups.

Participants will:

* Engage in nine structured modules of either internet-based CBT or sCBT
* Complete self-reported questionnaires on gambling severity and secondary symptoms at eight time points
* Have the option for up to three additional support sessions with a psychologist

DETAILED DESCRIPTION:
PROJECT GROUP: Anna Westh Stenbro (Psychologist, MSc.); Lisbeth Frostholm (Professor, Psychologist, MSc., Ph.D.); David Hodgins (Professor, Psychologist, MSc., Ph.D.)

The trial will be conducted by the research group at the Research Clinic for Gambling Disorder, based at Aarhus University Hospital, Denmark. The clinic was established in 2007 and offers assessment and specialized treatment to patients with GD.

MEASUREMENTS:

Self-reported data from the participants are collected at seven time points: At baseline (T1), randomisation (T2), three time points mid-treatment (T3, T4, T5), end-of-treatment (T6) and at 3-month follow-up (T7, primary endpoint). Due to different treatment durations in the two arms, an additional measurement point (T7b) is added to control for the effect of time for participants in the SF group, at the time point when participants in the sCBT group complete the 3-month follow-up (week 30). At T6, all participants will be invited to participate in a 12-month follow-up study (T8).

During treatment, therapists register the length, and themes, of phone conversations and face-to-face sessions in SpilleFri and equally the length and overall themes of sessions in the sCBT arm. In both arms, therapists register involvement of concerned significant others in treatment sessions. In the sCBT arm, therapist register manual fidelity and covered intervention topics after each session. Deviations are described. At the end of the treatment course, the therapists evaluate participant engagement and treatment effect (CGI-I).

For a detailed list of the measures and measurement time points included, see the section "Outcome measures".

RANDOMIZATION:

Included patients will be randomized to SF or sCBT in a 1:1 ratio. Randomization takes place immediately following the inclusion conference. A member of the research group will perform the randomization using the randomization module in the online data collection program, REDCap. When the randomization module is activated, REDCap automatically and randomly assigns participants to one of the predefined study groups in randomization blocks randomly ranging between 8 and 12. All research group members and clinicians are blinded to the current randomization block size.

POWER CALCULATION:

Sample size estimation was done using simulation of mixed linear models in Stata version 17. The relative effects of SF and sCBT will be analysed using a pre-set non-inferiority margin, determining the margin within which SF can be less effective than sCBT without being declared clinically inferior to the standard treatment. Within this margin, any difference in effect will represent a clinically unimportant loss of effect.

Simulation parameters were informed by 1) previous clinical data from the RCGD on reduction in NODS for patients given sCBT and 2) reduction in NODS for patients in the SF feasibility study. Assuming baseline-EOT-FU trajectory in NODS-score of 7-1-1 in individual CBT condition and 7-2-2 in SF condition, power of .80 was reached for 100 patients (50 in each condition). To account for dropout and attrition, a sample size of 150 is ideal.

ANALYSIS:

The hypothesized non-inferiority of SF compared to individual CBT as measured by NODS will be analysed using 2-level mixed linear models with random intercept - i.e., repeated measures nested within patients. REML estimation will be employed. Model-predicted mean change in NODS from baseline to FU is estimated in both CBT and SF condition, and a 95% confidence interval for the difference in change, i.e., ΔCBT-ΔSF, is calculated. The null-hypothesis of inferiority is rejected if the upper bound of this confidence interval is greater than the inferiority bound defined to be -2 NODS-scale points, i.e., SF leads to a change in NODS not more than 2 points less than CBT. The inferiority bound was decided based on clinical experience from RCGD, judging how large a difference in NODS that is clinically visible.

Results will be analysed and reported according to the CONSORT statement. A statistician is continuously involved in the project.

ELIGIBILITY:
Inclusion Criteria:

To be included patients should:

* fulfil diagnostic criteria for GD (DSM-5).
* score 4 points or more on the National Opinion Research Centre Screen for Gambling Problems (NODS).
* be able to read, write, and speak Danish.
* have IT skills and access to the internet and a computer, smartphone, and/or tablet.

Exclusion Criteria:

Patients are excluded from participation if they:

* present with severe comorbid somatic disease, cognitive deficits, severe trauma, and/or psychiatric disorder (e.g. depression, bipolar disorder, substance abuse, ADHD) that is insufficiently treated at the time of assessment and/or is evaluated to constitute a barrier for engaging in or benefitting from treatment.
* are not willing to engage in internet-delivered treatment or face-to-face cognitive behavioural therapy.
* do not provide informed consent.
* are in risk of suicide (indicated by clear intent and/or plans).
* have previously received treatment via or had access to the SpilleFri platform.
* seek treatment as part of an imminent legal case.
* only fulfil diagnostic criteria for Gambling Disorder in relation to behaviour such as stock trading or buying and selling cryptocurrency.
* present with highly unstable social circumstances, which are considered to potentially pose a barrier to engaging in treatment (e.g., homelessness).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2025-02-24 (Actual); Primary Completion 2027-01 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Change in Gambling Problems Past Month as Assessed by The National Opinion Research Center DSM Screen for Gambling Problems (NODS) | Baseline, 12 weeks/18 weeks (post treatment SpilleFri/sCBT), 24 weeks/30 weeks (3 month FU SpilleFri/sCBT), 64 weeks/70 weeks (12 month FU SpilleFri/sCBT)
  Measured by Danish translation of The National Opinion Research Center Screen for Gambling Problems (NODS). 17 items with a minimum score of 0 and a maximum score of 10, with higher scores meaning more servere gambling problems. Self-report measure collected through a web-based questionnaire program. For the purpose of the study, the NODS is modified to assess the last month instead of the last year.

SECONDARY OUTCOMES:
Change in Gambling Symptoms past week as Assessed by Gambling Symptom Assessment Scale (G-SAS) | Baseline, during treatment (weeks 4, 7, 10), post (week 12/18), 3 month FU (week 24/30), 12 month FU (week 64/70)
  The Gambling-Symptom Assessment Scale (G-SAS) is a 12-item self-rated measure that is designed to assess gambling symptom severity and change during treatment. Each item is scored on a 4-point scale from 0-4 with 0 meaning no symptoms and 4 meaning extreme symptoms. The total maximum score is 48.
Change in Self-reported Gambling Net Loss past week as assessed by a single item | Baseline, during treatment (weeks 4, 7, 10), post (week 12/18), 3 month FU (week 24/30), 12 month FU (week 64/70)
  Estimated net loss past week. Single-item self-report measure collected through a web-based questionnaire program.
Overall health improvement | Post (week 12/18, clinician rating), 3 month FU (week 24/30, participant and clinician rating)
  Measured by the 5-point clinical global improvement scale (CGI). The CGI is measured by self-report (CGI_p) and by clinician rating (CGI_c). 1 item assessing overall improvement or worsening on a 5-point scale with a maximum score of 5 and a minimum score of 1, with higher scores meaning a better outcome. Self-report measure collected throguh a web-based questionnaire program.
Change in Symptoms of anxiety, depression, and psychological distress as Assessed by th SCL-90 | Baseline, post (week 12/18), 3 month FU (week 24/30), 12 month FU (week 64/70)
  Measured by 13 relevant subscores of the 92-item Danish version of the Symptom Checklist (SCL-92). All items are rated on 5point scales. Maximum and minimum scores for the items are respectively 20 and 4 for anxiety, 30 and 6 for depression, and 40 and 8 for general distress, with higher scores meaning worse outcomes, i.e. more symptoms. Self-report collected through a web-based questionnaire program.
Change in Overall Quality of Life and General Health Satisfaction as Assessed by the WHOQoL | Baseline, post (week 12/18), 3 month FU (week 24/30), 12 month FU (week 64/70)
  Overall quality of life and general health satisfaction is measured using two single-item subscales from the WHOQoL. Both items are scored on five-point Likert-scales with 1 indicating very poor quality of life/very low general health satisfaction, and 5 indicating best possible quality of life/health satisfaction.
Change in Quality of Current Romantic Relationship as Assessed by the DAS-4 | Baseline, post (week 12/18), 3 month FU (week 24/30), 12 month FU (week 64/70)
  For participants who indicate that they are in a committed romantic relationship at baseline, the Dyadic Adjustment Scale, Brief Version (DAS-4) is used to measure the quality of the current relationship.The DAS-4 consists of four items with a maximum score of 21, indicating a very high relationship quality, and a minimum score of 0.
Participant treatment expectancy and satisfaction as Assessed by the Experienced Treatment Credibility and Expectancy | Baseline and post (week 12/18)
  Measured by the credibility/expectancy questionnaire. 6 items rated on a 1-9 or a 0%-100% scale, depending upon the item. The scale yields a mean expectancy/satisfaction score, ranging from maximum 100 % to minimum 0 %, with higher scores meaning higher expectancy of/satisfaction with the treatment. Self- report collected through a web-based questionnaire program

OTHER OUTCOMES:
Gambling Motives as Assessed by the Gambling Motives Questionnaire-Financial (GMQ-F) | Baseline
  Measured by the Gambling Motives Questionnaire-Financial (GMQ-F). The scale is condensed by selecting the two items with the highest factor loadings from each subscale, resulting in a total of 8 items. The scale assesses four primary motives for gambling: coping, enhancement, social, and financial. Each gambling motive has a maximum score of 8 and a minimum score of 2, with higher scores meaning higher degree of endorsement of the motive. Respondents are categorized based on their primary gambling motives, i.e. the gambling motive that is rated with the highest score. Self-report measure collected through a web-based questionnaire program.
Gambling pathway subtype as Assessed by the Gambling Pathways Questionnaire, GPQ | Baseline
  Measured by the Gambling Pathways Questionnaire (GPQ). 48 items with a maximum score of 288 and a minimum score of 48. The scale assesses etiological risk factors for problem gambling and categorizes respondents into one of three etiological subtypes, based on which of the following categories are scored the highest: Behaviorally Conditioned, Emotionally Vulnerable, and Antisocial-Impulsive. Self-report measure collected through a web-based questionnaire program
Change in Maladaptive Gambling Cognitions as Assessed by the Gambling-Related Cognitions Scale | Baseline, during treatment (weeks 4, 7, 10), post (week 12/18), 3 month FU (week 24/30), 12 month FU (week 64/70)
  To measure maladaptive gambling cognitions and gambling related self-efficacy, a shortened version of the Gambling-Related Cognitions Scale (GRCS; Raylu & Oei, 2004) is used. The scale is condensed by selecting the two items with the highest factor loadings from each subscale, resulting in a total of 10 items. On each of the five subscales, maximum scores of 14 indicate servere maladaptive cognitions, and minimum scores of 2 indicate no maladaptive cognitions.
Change in Difficulties in Emotion Regulation as Assessed by the DERS-16 | Baseline, during treatment (weeks 4, 7, 10), post (week 12/18), 3 month FU (week 24/30), 12 month FU (week 64/70)
  To measure difficulties in emotion regulation, the Difficulties in Emotion Regulation Scale (DERS-16) is used. The DERS-16 consists of 16 five-point Likert-scale items, with maximum scores of 80 indicating servere difficulties and minimum scores of 16 indicating no difficulties.
Participant activity in treatment program: Number of logins | Collected during treatment (week 1 to week 12/18)
  Collected through logged data from the treatment program "SpilleFri"
Contact with therapist per patient | Therapist report collected at post (week 12/18). Logged data collected during treatment (week 1 to week 12/18)
  Collected through therapist report in web-based questionnaire and logged data from the treatment program "SpilleFri".
Participant activity in treatment program: Time of the day of logins | Collected during treatment (week 1 to week 12/18)
  Collected through logged data from the treatment program "SpilleFri"
Participant activity in treatment program: Number of messages written to and received from therapists | Collected during treatment (week 1 to week 12/18)
  Collected through logged data from the treatment program "SpilleFri"
Participant activity in treatment program: Textual content written in exercises and messages | Collected during treatment (week 1 to week 12/18)
  Collected through logged data from the treatment program "SpilleFri"
Participant activity in treatment program: Total time spent in the program, on each module, on each page | Collected during treatment (week 1 to week 12/18)
  Collected through logged data from the treatment program "SpilleFri"

CONTACTS AND LOCATIONS:
Locations (1):
- Aarhus University Hospital, Aarhus, Denmark, Denmark

IPD SHARING:
Plan to Share IPD: No
To protect participant anonymity, individual participant data (IPD) will not be shared. Instead, aggregate data will be shared in an anonymized form.